CLINICAL TRIAL: NCT01284998
Title: Short Term Follow-up of Patent Implanted With the B-BOP Lock Plate
Status: Completed | Type: Observational
Sponsor: Integra LifeSciences Services (Industry)
Responsible Party: Sponsor
Other Study IDs: RECON-EMEA-07
Record Dates: First submitted 2011-01-26; First posted 2011-01-27 (Estimated); Last update posted 2014-09-11 (Estimated); Status verified 2014-09

CONDITIONS: Hallux Valgus; Hallux Varus; Vicious Callus on M1
Keywords: forefoot deformities; basal osteotomy
MeSH Terms: conditions — Hallux Valgus; Hallux Varus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- B-BOP lock: Subjects who needs a fixation of osteotomy of the basis of the first metatarsal and for whose surgeon has recommended that a B-BOP® Lock plate from INTEGRA be implanted can be enrolled in this study

SUMMARY:
In case of deformities of the forefoot (Hallux-valgus, Hallux-varus), the basal osteotomy may be more indicated than the distal osteotomy as it allows to achieve a greater degree of correction.

However, weight bearing forces on the head of the first metatarsal acting at a distance from the osteotomy site subject the construct to an important dorsiflexion stress. Fixation strength being the important consideration led to design the B-BOP® Lock plate, specifically dedicated to basal osteotomy of the first metatarsal, with the following characteristics:

* plantar positioning to obtain the best stability and resistance while reducing the implant bulkiness;
* anatomical shape adapted to the plantar curve of the first metatarsal. Taking advantages of the most appropriated anatomical site to implant the B-BOP® Lock plate directly on tension, it offers an innovative and unique basal osteotomy fixation solution.

The B-BOP® Lock osteosynthesis plate benefits now of the Surfix locking screws technology.

The purpose of this study is to collect and publish data from several centers, several users.

ELIGIBILITY:
Inclusion Criteria:

* Subject of either gender who needs a fixation of osteotomy of the basis of the first metatarsal for whose surgeon has recommended that a B-BOP® Lock plate from INTEGRA be implanted can be enrolled in this study.
* Age ≥ 18 years
* Have willingness to give his/her data transfer authorisation

Exclusion Criteria:

* Contraindication of the implantation of the B-BOP Lock plate
* History of prior mental illness or patient demonstrates that their mental capacity may interfere with their ability to follow the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who need a fixation of osteotomy of the basis of the first metatarsal.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2009-06; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Rate of device related complications. | 12 months
Iprovement of American Orthopaedic Foot and Ankle Society Hallux Metatarsophalangeal-lnterphalangeal Scale (AOFAS HMIS) score | 12 months

SECONDARY OUTCOMES:
X rays evaluation | 3 and12 months
Pain using a visual analog scale | 3 and 12 months
Function assessment | 3 and 12 Months
Clinical assessment | 3 and 12 months

CONTACTS AND LOCATIONS:
Locations (3):
- Clinique du Mont Louis, Paris, France
- Centre Hospitalier universitaire Notre Dame de secours, Byblos, Lebanon
- Wrexham Maelor Hospital, Wrexham, United Kingdom